CLINICAL TRIAL: NCT06566521
Title: Effect of Thoracic Paravertebral Block on Analgesia and the Quality of Recovery Following Daytime Laparoscopic Partial Adrenalectomy
Brief Title: Thoracic Paravertebral Block in Daytime Laparoscopic Partial Adrenalectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YXLL-2024-144
Record Dates: First submitted 2024-08-18; First posted 2024-08-22 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Laparoscopic Adrenalectomy; Day Surgery
Keywords: laparoscopic partial adrenalectomy; thoracic paravertebral block; daytime mode; analgesia; recovery quality
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPVB group (Experimental): After surgery and before extubation, the patient was positioned in an upper lateral position on the affected side. For patients in the TPVB group, an ultrasound high-frequency linear array probe was used to perform a mid-sagittal scan at the T8-9 spinous process interspace on the affected side. The probe was moved to visualize the T8-9 transverse process and pleura. Using the out-of-plane needling technique, the needle was inserted between the costotransverse ligament and the pleura in the paravertebral space adjacent to the thoracic vertebra. After confirmation of no blood or cerebrospinal fluid return, 30 mL of 0.5% ropivacaine hydrochloride was injected. Under ultrasound guidance, the spread of the medication and downdraft of the pleura could be observed.
  Interventions: Procedure: thoracic paravertebral block
- control group (No Intervention): The patients in the control group did not undergo the nerve block procedure.

INTERVENTIONS:
Procedure: thoracic paravertebral block — After surgery and before extubation, the patient was positioned in an upper lateral position on the affected side. For patients in the TPVB group, an ultrasound high-frequency linear array probe was used to perform a mid-sagittal scan at the T8-9 spinous process interspace on the affected side. The probe was moved to visualize the T8-9 transverse process and pleura. Using the out-of-plane needling technique, the needle was inserted between the costotransverse ligament and the pleura in the paravertebral space adjacent to the thoracic vertebra. After confirmation of no blood or cerebrospinal fluid return, 30 mL of 0.5% ropivacaine hydrochloride was injected. Under ultrasound guidance, the spread of the medication and downdraft of the pleura could be observed.
  Arms: TPVB group

SUMMARY:
Day surgery refers to the entire diagnostic and therapeutic process completed within 24-48 h, including patient admission, surgery, and discharge. Research by Shariq et al suggested that daytime laparoscopic adrenalectomy was a safe and effective alternative to traditional inpatient treatment. Li et al demonstrated that daytime surgery for laparoscopic partial adrenalectomy could reduce hospital stays, lower medical costs, and optimize healthcare resource utilization.

The day surgery has put forward higher requirements for the management of perioperative anesthesia, in which the postoperative multimodal analgesia is particularly important.Thoracic paravertebral block (TPVB) is a regional block technique in which local anaesthetics can be injected into paravertebral space to block the ipsilateral sympathetic and somatosensory nerves. TPVB single point injection can achieve sensory block of 3-6 spinal ganglia on one side, with minimal impact on respiratory, gastrointestinal and bladder function. Especially, TPVB does not affect motor nerve, which enable patients to perform painless functional exercise shortly after surgery, promote rapid recovery, and enhance satisfaction and comfort.

A large number of previous studies have shown that TPVB had become increasingly popular for postoperative analgesia after thoracic or breast surgery. However, to our knowledge, few studies to date have investigated the application of TPVB in daytime adrenal surgery. Therefore, we conducted this randomized clinical trial to examine the effect of TPVB on postoperative analgesia and the quality of recovery in patients following daytime laparoscopic partial adrenalectomy.

DETAILED DESCRIPTION:
1. Study purpose

   To investigate the impact of thoracic paravertebral block for postoperative analgesia and quality of recovery following daytime laparoscopic partial adrenalectomy.
2. Study design

   2.1. Type of the study

   The research is a single-center, double-blind, randomized-controlled clinical trial.

   2.2 Sample size calculation

   The estimated sample size was calculated using SPSS Statistics, version 26.0 ((IBM Corp), and this was based on our preliminary study, in which the scores of the QoR-15 scale (points, mean ± standard deviation) of the control group and the TPVB group at 24 hours postoperatively were 116.2±6.7 and 124.3±8.8, respectively. The test level α was set to 0.05, the test power 1-β was set to 0.90. The sample size was determined to be 28 patients in each group. Considering a dropout rate of approximately 20%, 35 individuals were included in each arm of this trial.

   2.3 Randomization and blinding

   Patients were randomly assigned in a 1:1 ratio into 2 groups, the control group or the TPVB group via centrally computer-generated group randomization. Immediately after the surgery, a sealed opaque envelope containing the patient group assignment was opened by an experienced anesthesiologist in charge. TPVB was performed by the same anesthesiologist for the patients in the TPVB group, while the patien in the control group did not receive nerve blockade.

   Participants in the control and TPVB groups were kept blinded to their group assignment. This study involved researchers who conducted the postoperative follow-up and evaluation (blinded) and researchers who administered the treatment (unblinded). The unblinded researchers who administered the interventions were not involved in the evaluation of the postoperative outcomes.

   2.4 Intervention protocol

   After surgery and before extubation, the patient was positioned in an upper lateral position on the affected side. For patients in the TPVB group, an ultrasound high-frequency linear array probe was used to perform a mid-sagittal scan at the T8-9 spinous process interspace on the affected side. The probe was moved to visualize the T8-9 transverse process and pleura. Using the out-of-plane needling technique, the needle was inserted between the costotransverse ligament and the pleura in the paravertebral space adjacent to the thoracic vertebra. After confirmation of no blood or cerebrospinal fluid return, 30 mL of 0.5% ropivacaine hydrochloride was injected. Under ultrasound guidance, the spread of the medication and downdraft of the pleura could be observed. The patients in the control group did not undergo the nerve block procedure.
3. Adverse events

   Including postoperative nausea and vomiting, as well as postoperative agitation and nerve block- related complications, such as bleeding, hematoma, pneumothorax, or nerve injury
4. Quality control

   All research data, both in paper and electronic formats, will be kept for at least 5 years. If readers have any questions after the article's publication, they may contact the corresponding author for access to the original data. Patient information will remain anonymous, including name, ID number and telephone number. All data related to enrolled patients collected during the study period of this project will be archived and safeguarded, and all study members and study sponsors are asked to keep subject information confidential. The study protocol will be reviewed and revised by statistical experts. Investigators will adhere to pre-defined standard operating procedures, encompassing patient screening, follow-up standardization, result assessment, and data management. The Ethics Committee of Shanxi Bethune Hospital will review the trial every six months.
5. Statistical analysis

Statistical analysis was performed using SPSS Statistics, version 26.0. Normally distributed continuous variables were presented as mean (SD) values, and intergroup comparisons used independent-sample t-test. Nonnormally distributed variables were presented as median (IQR) values, and intergroup comparisons were determined using the Mann-Whitney test. Categorical variables were expressed as frequencies and percentages, and these were compared using either the χ2 test or the Fisher exact test. A P<0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to70 years
* Body Mass Index (BMI) 18.5 to 30 kg/m²
* American Society of Anesthesiologists (ASA) grade I to II classification
* unilateral non-functional adrenal adenoma with a tumor diameter greater than 20mm

Exclusion Criteria:

* Patients with peripheral nervous system disease
* Patients with spinal deformity or surgery
* Patients with puncture site infection or coagulation abnormalities
* Patients with history of postoperative nausea and vomiting or allergy to local anesthetics
* Patients with unstable mental illness or refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | 24 and 48 hours postoperatively
  quality of recovery, measured using the 15-item Quality of Recovery questionnaire (QoR-15), It ranges from 0 to 150, with a higher score indicating a better quality of recovery

SECONDARY OUTCOMES:
pain scores at rest and during coughing | 1, 6, 12, 24, and 48 hours after surgery
  pain scores, measured using the Visual Analog Scale(0 points indicated no pain, a score <4 indicated mild pain; a 4-7 score indicated moderate pain, a score >7 points indicated severe pain, and a score of 10 indicated unbearably severe pain)
Opioid consumption | 48 hours postoperatively
  The total amount of sufentanil used in the PCA pump within the initial 48 h postoperatively
Rate of remedial analgesia | 48 hours postoperatively
  The rate of remedial analgesia 48 hours postoperatively
Postoperative gastrointestinal function outcomes | 12, 24, and 48 hours after suegery
  I-FEED scores(an I-FEED scores of 0-2 indicates postoperative gastrointestinal normality, 3-5 indicates postoperative gastrointestinal intolerance, and ≥6 indicates postoperative gastrointestinal dysfunction)
Times to first flatus and defecation | 48 hours postoperatively
  The time of first flatus and defecation within 48h after operation was measured by hour

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Wen Zhang, MD, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China